CLINICAL TRIAL: NCT01752764
Title: Assessment of the Relative Increase in Bioavailability of (Non-) Nutrients From a Mixed Salad by Adding Fat Containing Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FDS-DRS-0573
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Experimental): Test product: Salad with high dosage fat
  Interventions: Other: Test product: Salad with a high dosage fat; Other: Control product: Salad with low dosage fat
- Control product (Other): Control product: Salad with low dosage fat
  Interventions: Other: Test product: Salad with a high dosage fat; Other: Control product: Salad with low dosage fat

INTERVENTIONS:
Other: Test product: Salad with a high dosage fat
Other: Control product: Salad with low dosage fat

SUMMARY:
The hypothesis will be tested that fat can also increase absorption of (non)-nutrients from a salad. Therefore we designed the current study to show an increase in relative absorption (bioavailability) of (non-) nutrients from a mixed salad by adding fat containing dressing.

ELIGIBILITY:
Main inclusion Criteria:

* Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2.
* Apparently healthy: no medical conditions, no use of prescribed or over the counter drugs, which might affect study measurements (as judged by study physician)
* Haemoglobin within normal reference range as judged by the study physician.
* Total cholesterol, LDL cholesterol, HDL cholesterol and fasting triglycerides within the normal reference range, as judged by the study physician.

Main exclusion Criteria:

* Reported use of any medically- or self-prescribed diet at the moment of screening, or the intention to use any kind of diet in the period between screening and the end of the study.
* Reported weight loss or gain ≥ 10 % of bodyweight during a period of six months before screening.
* A known food allergy or intolerance.
* A dislike to the foods supplied during the study.
* Use of vitamins or supplements enriched with carotenoid and/or vitamin A and/of vitamin K.
* Known hypothyroidism or hyperthyroidism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC in nmol/l*h) of (non) nutrients | July 2013
  Area under the curve (AUC in nmol/l*h) of (non) nutrients. The AUCs are constructed from (non-) nutrient levels measured in plasma chylomicrons at the selected time-points. The size of the areas under the curves will be compared between the test and control dressing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Raul C. Maranhão, M.D, Ph.D., Principal Investigator — Head Professor of Clinical Biochemistry, Faculty of Pharmaceutical Sciences Director, Lipid Metabolism Laboratory
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo / Incor HC FM USP, São Paulo, Av. Dr. Enéas de Carvalho Aguiar, 44, Brazil